CLINICAL TRIAL: NCT05565391
Title: Comparative Effectiveness of Elranatamab (PF 06863135) in Clinical Study C1071003 Versus Standard of Care (SOC) in Real-World (RW) External Control Arms in Patients With Triple-Class Refractory (TCR) Multiple Myeloma (MM)
Brief Title: A Study to Learn About the Medicine (Called Elranatamab) in People With Relapsed Refractory Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C1071024
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Results first posted 2024-04-22 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Multiple Myeloma; relapsed Multiple Myeloma; refractory Multiple Myeloma; PF-06863135; BCMA; bispecific; bispecific antibody; BCMA-CD3 bispecific; Elranatamab; MagnetisMM-3
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Elranatamab: Patients treated with elranatamab from the MagnetisMM-3 trial
  Interventions: Drug: Elranatamab
- Standard of care: Patients treated with standard-of-care therapies from real-world data sources
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Elranatamab — BCMA-CD3 bispecific antibody
  Groups: Elranatamab
Drug: Standard of care — Standard of care
  Groups: Standard of care

SUMMARY:
This study is to understand how well elranatamab (PF-06863135) may be used for relapsed refractory multiple myeloma (RRMM). Sometimes MM might improve at first, but then gets resistant to the treatment and starts growing again (known as relapsed refractory). This study medicine will be compared with standard-of-care (SOC) therapies used in real-world clinical practice. For people receiving elranatamab, we will use data from the phase 2 clinical trial (MagnetisMM-3). We will also use data from two real-world databases, representing the SOC in clinical practice. This study does not seek any participants for enrollment. We will compare the experiences of people receiving elranatamab to people receiving SOC therapies. This way, it will help us to know how well elranatamab can be used for RRMM treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older at index date
* Diagnosis of MM
* Measurable disease according to IMWG criteria
* ECOG performance status ≤2
* Refractory to at least 1 proteasome inhibitor, 1 immunomodulatory drug, and 1 anti-CD38 treatment (ie, triple-class refractory [TCR])
* At least 1 treatment following their TCR eligibility

Exclusion Criteria:

* Acute plasma cell leukemia
* Amyloidosis
* Smoldering MM
* Stem cell transplant within 12 weeks of index or active graft versus host disease (GVHD)
* Active malignancy within 3 years before index, except for basal cell or squamous cell skin cancer or carcinoma in situ
* Administration with an investigational drug within 30 days prior to index

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with elranatamab will come from the MagnetisMM-3 trial. Patients treated with the standard-of-care therapies will come from electronic health record databases in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 508 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This retrospective cohort study included triple-class refractory (TCR) multiple myeloma (MM) participants who initiated elranatamab in study C1071003 (NCT04649359) and 2 cohorts of real-world (RW) TCR MM participants who initiated standard of care (SOC) treatment identified from Flatiron Health and COTA databases as external control arms for Study C1071003.
Pre-assignment Details: Index date was defined as the date of initiation of the first regimen after TCR MM eligibility. Only participants with an index date between 16-Nov-2015 and 31-Mar-2022 were selected. Participants were observed from the index date to the earliest of death, or the latest available participants record, whichever occurred first.
Groups:
- Study C1071003 Cohort A: Participants with TCR MM who initiated elranatamab (PF-06863135) following TCR eligibility in study C1071003 (NCT04649359) were included.
- COTA Cohort: Participants with RW TCR MM who initiated standard of care treatment following TCR eligibility between 16-Nov-2015 and 31-Mar-2022 identified from COTA database were included.
- Flatiron Health Cohort: Participants with RW TCR MM who initiated standard of care treatment following TCR eligibility between 16-Nov-2015 and 31-Mar-2022 identified from Flatiron Health database were included.
Period: Overall Study
Arm/Group | Study C1071003 Cohort A | COTA Cohort | Flatiron Health Cohort
Started | 123 | 233 | 152
Completed | 123 | 233 | 152
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants from study C1071003 (Cohort A) and RW participants identified from COTA and Flatiron Health databases were included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Study C1071003 Cohort A | COTA Cohort | Flatiron Health Cohort | Total
Number analyzed (Participants) | 123 | 233 | 152 | 508
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  >18 years | 123 | 233 | 152 | 508
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 107 | 72 | 234
  Male | 68 | 126 | 80 | 274
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 72 | 170 | 102 | 344
  Non-white | 51 | 63 | 50 | 164

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)-Unweighted Analysis
Description: ORR was the percentage of participants with objective response (OR) per IMWG criteria. For the analysis set of participants from Study C1071003 and COTA, OR was partial response (PR) or better (stringent complete response [sCR]+complete response [CR]+very good partial response [VGPR]+PR). For Study C1071003 and Flatiron Health, OR was PR or better (at least VGPR+PR). sCR: CR & normal serum free light chain (sFLC) ratio & absence of clonal cells in BMB/BMA by IH, IF, or flow cytometry. CR: negative immunofixation on serum & urine, disappearance of any soft tissue plasmacytoma & <5% plasma cells in BMA, if measured by sFLC only, preceding criteria + normal sFLC ratio. VGPR: Serum & urine M-protein detectable by immunofixation but not on electrophoresis; or >=90% reduction in serum & urine M-protein level <100mg/24h. PR: >=50% reduction in serum M-protein & reduction in 24h urinary M-protein by >=90% or <200 mg/24h. Clopper-Pearson two-sided 95% exact confidence intervals were estimated.
Time Frame: From index date until first documentation of progression, death, or the start of new anticancer therapy (median follow-up of 10.4 months for study C1071003 cohort A, 8.8 months and 7.7 months for COTA and Flatiron Health cohorts)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Study C1071003 Cohort A | COTA Cohort | Flatiron Health Cohort
Number analyzed (Participants) | 123 | 233 | 152
Percentage of participants | 61.0 [51.8 to 69.6] | 31.3 [25.4 to 37.7] | 30.3 [23.1 to 38.2]
Statistical Analysis 1: Comparison: Study C1071003 Cohort A vs COTA Cohort; Test type: Other; p < .0001, Log-binomial regression model; Risk Ratio (RR) = 1.95, 95% CI 2-sided [1.54 to 2.47] — Unweighted RRs were estimated using a log-binomial regression model with Wald confidence intervals
Statistical Analysis 2: Comparison: Study C1071003 Cohort A vs Flatiron Health Cohort; Test type: Other; p < .0001, Log-binomial regression model; Risk Ratio (RR) = 2.01, 95% CI 2-sided [1.52 to 2.67] — Unweighted RRs were estimated using a log-binomial regression model with Wald confidence intervals

2. Primary Outcome: Objective Response Rate-Comparison Between Elranatamab in Study C1071003 Cohort A and COTA Cohort Using Inverse Probability of Treatment Weights (IPTW) Analysis
Description: ORR was the percentage of participants with an OR per IMWG criteria. For the analysis set of participants from Study C1071003 and COTA, the OR was defined as PR or better (sCR + CR + VGPR + PR). For Study C1071003 and Flatiron Health, OR was defined as PR or better (at least VGPR + PR). sCR: CR & normal serum free light chain (sFLC) ratio & absence of clonal cells in BMB/BMA by IH, IF, or flow cytometry. CR: negative immunofixation on serum & urine, disappearance of any soft tissue plasmacytoma & <5% plasma cells in BMA, if measured by sFLC only, preceding criteria + normal sFLC ratio. VGPR: Serum & urine M-protein detectable by immunofixation but not on electrophoresis; or >=90% reduction in serum & urine M-protein level <100mg/24h. PR: >=50% reduction in serum M-protein & reduction in 24h urinary M-protein by >=90% or <200 mg/24h. Analysis was performed using IPTW method to balance participant characteristics among reporting groups.
Time Frame: as for outcome 1
Population: Eligible participants from study C1071003 (Cohort A) and RW participants identified from COTA and Flatiron Health databases were included. Here, "Overall Number of Participants Analyzed" is the number of participants after application of IPTW method to raw numbers and is different from the actual participants included in the reporting arm.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Study C1071003 Cohort A | COTA Cohort
Number analyzed (Participants) | 123 | 213
Percentage of participants | 75.7 [65.6 to 87.4] | 34.2 [27.2 to 43.0]
Statistical Analysis 1: Comparison: Study C1071003 Cohort A vs COTA Cohort; Test type: Other; p < .0001, Log-binomial regression model; Risk Ratio (RR) = 2.22, 95% CI 2-sided [1.69 to 2.90] — Risk ratio was estimated using a log-binomial regression model and confidence interval was estimated using robust error variance

3. Primary Outcome: Objective Response Rate-Comparison Between Elranatamab in Study C1071003 Cohort A and Flatiron Health Cohort Using IPTW Analysis
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Study C1071003 Cohort A | Flatiron Health Cohort
Number analyzed (Participants) | 122 | 149
Percentage of participants | 56.0 [41.1 to 76.2] | 31.3 [19.4 to 50.4]
Statistical Analysis 1: Comparison: Study C1071003 Cohort A vs Flatiron Health Cohort; Test type: Other; p = 0.0447, Log-binomial regression model; Risk Ratio (RR) = 1.79, 95% CI 2-sided [1.01 to 3.15] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Time to Response (TTR)-Unweighted Analysis
Description: TTR was defined as the time from the index date to the first documentation of OR. No censoring was performed. OR is defined as having a best overall response (BOR) of confirmed sCR, CR, VGPR or PR per IMWG criteria.
Time Frame: From index date to date of first documentation of OR (median follow-up of 10.4 months for study C1071003 cohort A, 8.8 months and 7.7 months for COTA and Flatiron Health cohorts)
Population: Eligible participants from study C1071003 (Cohort A) and RW participants identified from COTA and Flatiron Health databases were included. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Study C1071003 Cohort A | COTA Cohort | Flatiron Health Cohort
Number analyzed (Participants) | 75 | 73 | 46
Months | 1.22 [0.99 to 2.00] | 1.38 [0.82 to 2.79] | 1.87 [0.95 to 2.69]
Statistical Analysis 1: Comparison: Study C1071003 Cohort A vs COTA Cohort; Test type: Other; p = 0.4241, Quantile regression
Statistical Analysis 2: Comparison: Study C1071003 Cohort A vs Flatiron Health Cohort; Test type: Other; p = 0.0281, Quantile regression

5. Secondary Outcome: Time to Response (TTR)-Comparison Between Elranatamab in Study C1071003 Cohort A and COTA Cohort Using IPTW Analysis
Description: TTR was defined as the time from the index date to the first documentation of OR. OR is defined as having a best overall response (BOR) of confirmed sCR, CR, VGPR or PR per IMWG criteria. Analysis was performed using IPTW method to balance participant characteristics among reporting groups.
Time Frame: as for outcome 4
Population: Eligible participants from study C1071003 (Cohort A) and RW participants identified from COTA and Flatiron Health databases were included. Here, "Overall Number of Participants Analyzed" is the number of participants after application of IPTW method to raw numbers.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Study C1071003 Cohort A | COTA Cohort
Number analyzed (Participants) | 76 | 68
months | 1.25 [0.99 to 2.10] | 1.18 [0.82 to 1.87]
Statistical Analysis 1: Comparison: Study C1071003 Cohort A vs COTA Cohort; Test type: Other; p = 0.7682, Quantile regression

6. Secondary Outcome: Time to Response-Comparison Between Elranatamab in Study C1071003 Cohort A and Flatiron Health Cohort Using IPTW Analysis
Description: as for outcome 5
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Study C1071003 Cohort A | Flatiron Health Cohort
Number analyzed (Participants) | 74 | 43
Months | 1.15 [0.99 to 2.00] | 1.87 [0.95 to 2.10]
Statistical Analysis 1: Comparison: Study C1071003 Cohort A vs Flatiron Health Cohort; Test type: Other; p = 0.0326, Quantile regression

7. Secondary Outcome: Duration of Response (DOR)-Unweighted Analysis
Description: DOR was defined as the time from the first documentation of OR, until confirmed disease progression (PD) per IMWG criteria, or death due to any cause, whichever occurred first. PD= increase of >=25% from lowest value in >=1 of following (serum M-protein [absolute increase >=0.5g/dL]; serum M-protein increase >=1g/dL [when lowest M-protein >=5g/dL]; and urine M-protein [absolute increase >=200mg/24h]).
Time Frame: From first documentation of OR until confirmed PD or death due to any cause or censoring date (median follow-up of 10.4 months for study C1071003 cohort A, 8.8 months and 7.7 months for COTA and Flatiron Health cohorts)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Study C1071003 Cohort A | COTA Cohort | Flatiron Health Cohort
Number analyzed (Participants) | 75 | 73 | 46
Months | NA [11.99 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 4.37 [2.86 to 8.05] | 7.16 [4.99 to 13.60]
Statistical Analysis 1: Comparison: Study C1071003 Cohort A vs COTA Cohort; Test type: Other; p < .0001, Cox proportional hazard model; Hazard Ratio (HR) = 0.17, 95% CI 2-sided [0.09 to 0.31] — Hazard ratio was estimated using unadjusted Cox proportional hazard model
Statistical Analysis 2: Comparison: Study C1071003 Cohort A vs Flatiron Health Cohort; Test type: Other; p < .0001, Cox proportional hazard model; Hazard Ratio (HR) = 0.22, 95% CI 2-sided [0.11 to 0.43] — Hazard ratio was estimated using unadjusted Cox proportional hazard model

8. Secondary Outcome: Duration of Response-Comparison Between Elranatamab in Study C1071003 Cohort A and COTA Cohort Using IPTW Analysis
Description: DOR was defined as the time from the first documentation of OR, until confirmed disease progression (PD) per IMWG criteria, or death due to any cause, whichever occurred first. PD= increase of >=25% from lowest value in >=1 of following (serum M-protein [absolute increase >=0.5g/dL]; serum M-protein increase >=1g/dL [when lowest M-protein >=5g/dL]; and urine M-protein [absolute increase >=200mg/24h]). Median and 95% Confidence Interval (CI) reported in the descriptive section was determined using unweighted analysis.
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Study C1071003 Cohort A | COTA Cohort
Number analyzed (Participants) | 75 | 68
Months | NA [11.99 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 4.37 [2.86 to 8.05]
Statistical Analysis 1: Comparison: Study C1071003 Cohort A vs COTA Cohort; Test type: Other; p < .0001, Cox proportional hazard model; Hazard Ratio (HR) = 0.11, 95% CI 2-sided [0.06 to 0.22] — Hazard ratio was estimated using weighted Cox proportional hazard model and confidence interval was estimated using robust error variance

9. Secondary Outcome: Duration of Response-Comparison Between Elranatamab in Study C1071003 Cohort A and Flatiron Health Cohort Using IPTW Analysis
Description: as for outcome 8
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Study C1071003 Cohort A | Flatiron Health Cohort
Number analyzed (Participants) | 74 | 43
Months | NA [11.99 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 7.16 [4.99 to 13.60]
Statistical Analysis 1: Comparison: Study C1071003 Cohort A vs Flatiron Health Cohort; Test type: Other; p < .0001, Weighted Cox proportional hazard model; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.10 to 0.45] — [estimate comment as in outcome 8, analysis 1]

ADVERSE EVENTS:
Time Frame: Not applicable as safety data was not collected.
Description: This was a retrospective study and the data existed as structured data. In these data sources, individual participant data were not retrieved or validated, and it was not possible to link a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event could not be met, hence adverse events data were not collected and reported.
Groups:
- COTA Chohort: Participants with RW TCR MM who initiated standard of care treatment following TCR eligibility between 16-Nov-2015 and 31-Mar-2022 identified from COTA database were included.
Arm/Group | Study C1071003 Cohort A | COTA Chohort | Flatiron Health Cohort
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT05565391/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT05565391/SAP_001.pdf